CLINICAL TRIAL: NCT00580827
Title: Clinical Efficacy of Disulfiram in LAAM-Maintained Cocaine Abusers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: James Poling, Ph.D. / Research Scientist, Yale University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9811010624; R01DA013441 (NIH)
Record Dates: First submitted 2007-12-25; First posted 2007-12-27 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Cocaine-Related Disorder; Opiate Dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Disulfiram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo disulfiram (Placebo Comparator): placebo disulfiram (0 mg/day)
  Interventions: Drug: Placebo
- disulfiram 62.5 (Experimental): disulfiram at 62.5 mg/day
  Interventions: Drug: Disulfiram
- disulfiram 125 (Experimental): disulfiram at 125 mg/day
  Interventions: Drug: Disulfiram
- disulfiram 250 (Experimental): disulfiram at 250 mg/day
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Placebo — Matched placebo.
  Arms: placebo disulfiram
Drug: Disulfiram — disulfiram at 62.5 mg/day for 12 weeks.
  Arms: disulfiram 62.5
Drug: Disulfiram — Disulfiram at 125 mg/day for 12 weeks.
  Arms: disulfiram 125
Drug: Disulfiram — disulfiram at 250 mg/day for 12 weeks.
  Arms: disulfiram 250

SUMMARY:
This 18-week, randomized, double blind clinical trial provided treatment for 160 cocaine-dependent opioid addicts, aged 18-65 years. Participants were stabilized on LAAM maintenance during the first 4 weeks and cocaine use was assessed; participants were then stratified by level of cocaine use and randomly assigned to receive one of the following: placebo disulfiram (0 mg/day), disulfiram at 62.5 mg/day, disulfiram at 125 mg/day, or disulfiram at 250 mg/day. During induction onto LAAM, participants were administered increasing doses of LAAM plus placebo disulfiram on a thrice-weekly basis until maintenance doses of LAAM are attained. At the beginning of week 5, participants received LAAM plus disulfiram or placebo disulfiram according to their randomized assignments, and were maintained on these agents through week 16. At the end of the study, participants underwent detoxification from LAAM and active/placebo medication over a 4- to 6-week period. All participants received weekly 1-hour psychotherapy (Cognitive Behavioral Treatment) with experienced clinicians specifically trained to deliver the therapy and who received ongoing supervision. The primary outcomes were retention and reduction in opioid and cocaine use, as assessed by self-report and confirmed by thrice-weekly urinalyses. Secondary outcomes included reductions in other illicit drug and alcohol use, as well as improvements in psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years.
* Are not currently enrolled in treatment.
* Participants must demonstrate opioid dependence, as evidenced by documentation of prior opioid agonist maintenance and/or have signs of withdrawal upon administration of naloxone (<0.8 mg, i.m.), and an opioid-positive urine screen.
* Participants also must be current users of cocaine with self-reported use of > 7 gm during the preceding 12 months, self-reported use of > 1 time/week in at least one month preceding study entry, and cocaine-positive urine screen.
* Participants must fulfill DSM-IV criteria for opioid and cocaine dependence.

Exclusion Criteria:

* current diagnosis of other drug or alcohol physical dependence (other than opiates, cocaine or tobacco)
* significant medical conditions such as abnormal liver function (with laboratory findings greater than three times normal).
* active hepatitis; hypertension; a current cardiac condition or high risk of cardiovascular disease; seizure disorders; or another significant underlying medical condition which would contraindicate disulfiram or LAAM treatment.
* meets DSM-IV psychiatric classifications for schizophrenia, bipolar disorder, or other psychotic disorders; exhibiting current suicidality or homicidality; current use of a prescribed psychotropic medication that cannot be discontinued.
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2003-09; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Reductions in cocaine use as measured by urine toxicology and self-report | 14 weeks

SECONDARY OUTCOMES:
Predictors of treatment efficacy using DBH genotyping for disulfiram will be tested. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Poling, Ph.D., Principal Investigator — Yale University
Locations (1):
- West Haven VA, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Traccis F, Minozzi S, Trogu E, Vacca R, Vecchi S, Pani PP, Agabio R. Disulfiram for the treatment of cocaine dependence. Cochrane Database Syst Rev. 2024 Jan 5;1(1):CD007024. doi: 10.1002/14651858.CD007024.pub3. PMID 38180268